Achieving Competitive
Customized
Employment through
Specialized Services Veterans: ACCESSVETS

NCT04832802

February 20, 2024

## **SCRIPT (SCREENING & VERBAL CONSENT) VETERAN**

| Introduction: |
|---|
| Hello, my name is []. I am a member of the research team at James A Haley Veterans Hospital. |
| We are contacting you because you may qualify to participate in a research study that aims to help Veterans with Spinal Cord Injuries find meaningful employment. You may have heard about this study from VA staff, flyers, or social media. You may have also received a letter in the mail with study information. Would you mind if I took some time to talk with you about this study? |
| If at any time during this phone call, the Veteran answers "no" to a question, then state Thank you for your time. Please contact us at NUMBER if you have any questions about the study. Also, you can contact the VA Central IRB to confirm this is VA research: 1-877-254-3130. The information you have provided us today will not be used in the study and will be kept confidential. |
| <i>If the Veteran says "yes" then state</i> The study compares customized employment to supported employment programs. We hope the information from this study will improve VA employment services for Veterans with SCI. |
| If you participate, you will complete some questionnaires to tell us about yourself and your employment experiences. Then, you will be randomly selected (i.e., by chance) to work with a vocational specialist in an employment program for about 8 months to reach your employment goals. During the study, we will contact you to schedule 3 follow-up study visits to complete questionnaires that let us know how you are doing before, during, and after the employment program. You will receive payment (up to \$120.00) for time spent completing study activities. We anticipate that these surveys will take approximately 30 minutes to one hour to complete. Some participants will also be asked to participate in an open-ended audio-recorded interviews at three separate timepoints. You will receive payment for each interview (up to \$90). Is this a study that you'd be interested in if you meet the study criteria? |

## If the Veteran says "yes" then state...

Before you can enroll in the study, we need to ask you a few questions to determine if you meet certain requirements to participate. All information discussed will be confidential, except if you tell me you are going to hurt yourself or someone else or report abuse to a child, elder, or vulnerable person. You may refuse to answer any question and stop this interview at any time. Would you like to continue?

*If the Veteran says "ves" then state...* 

| If the veteral says yes then state |
|--------------------------------------------------------|
| Screening Questions |
| Inclusion Criteria |
| 1. Do you have any difficulties speaking or |
| understanding English? |
| 2. Are you 18 years of age or older? |
| 3. Do you want to find work in your community? |
| 4. Have you received or are you currently receiving VA |
| Individual Placement and Support services to find |
| employment (also called Compensated Work Therapy |
| Supported Employment)? |
| Exclusion Criteria |

| 1. | . Do you live more than two hours' drive from the VAMC? |
|---|---|
| 2. | 2. Do you have a progressive spinal cord disorder or a |
| | terminal diagnosis e.g., multiple sclerosis? |
| 3. | B. Do you have a moderate or severe traumatic brain injury? |
| 4. | I. Have you ever been treated for psychosis? Was your treatment within the last six months? Examples include schizophrenia and dementia |
| 5. | 5. Do you have an untreated substance abuse disorder? |
| 6. | 5. Do you have any visual, hearing, or cognitive impairments that prevent the ability to consent or participate in answering questionnaires or finding work? |

<u>If participants do not meet inclusion criteria the research team member could say:</u> I regret to inform you that you do not meet the requirements to participate in this study, but we appreciate your interest in this project. If you want more information about employment services, please talk to your treatment team about options at our VA.

*If participant meets inclusion/eligibility criteria (answered "yes" to inclusion criteria and "no" to exclusion criteria the research team member should say*: You meet the requirements to participate in the research study

If you are interested in participating, I can tell you more about the study now, or I can call you back when you have more time to talk. If you're not interested in the study, that's okay, you can tell me now and I won't contact you again.

*If participant is not interested in the study the research team member should say:* "Thank you very much for your time, goodbye."

| If participant is interested in the study: Is it okay to talk to you now, or may I call back at a better time?" |
|---|
| No (later). When would be a good day and time to call? |
| Yes (now). Go on with the script: |

At this time, I would like to review an information sheet about the study. You should have received a letter in the mail with a copy of this information sheet that outlines the study in more detail. If you do not have the information sheet available with you at this time, that's ok, I will mail a copy of it to you later for your reference.

Study staff reviews information sheet with Veteran and ensures that the Veteran has ample opportunity to discuss the information and ask questions.

Have you had enough time to review and think about this information?

| AGREEMENT TO PARTICIPATE I | N THE RESEARCH STUDY |
|---|---|
| Dr./Mr./Ms has explained the research study to you. You have been told of the risks or discomforts and possible benefits of the study. You have been told of other choices of treatment available to you. You have been given the chance to ask questions and obtain answers. | |
| Do you want to participate in this study? | Do you want to participate in this study? |
| NO | |
| YES | |
| Signature of Research Team Member O | btaining Consent |
| If no, say "Thank you, I really apprecia | te your taking the time to talk with me, goodbye." |
| If yes, go on with the script. | |
| experience with the employment program. These interviews are audio-recorded for typed out word for word, excluding any | articipants will be asked to do open-ended interviews about their m by a special member of the study team called a qualitative researcher accuracy. The study will then have the audio-recording transcribed, or identifying information. You will not be identified by name, and any will be removed from the transcript. Are you willing to be audiody? |
| YES, I agree to allow audio-record | ling of my study interview sessions. |
| NO, I do not agree to allow audio- | recording of my study interview sessions. |
| Signature of Research Team Member O | btaining Consent Date |
| | tion sheet for Veteran participants. It lists everything that we have formation for your records such as the name and contact information of he VA, Dr. Lisa Ottomanelli. |

Do you have questions for me at this time? If you later decide you have any questions, please contact Areana Cruz at 813-797-8969. Also, you can contact the VA Central IRB toll free at 1-877-254-3130 if you have any

Version 5

Version Date 10/24/2023

questions, complaints, or concerns about the study.

VA Central IRB Effective Date: February 20, 2024 At this point, we can set up a time for your first study visit. This visit will consist of a baseline questionnaire that let us know about yourself, your work history, and your goals. It will take about 30 minutes to an hour. Would you like to schedule that visit now?

## If the Veteran says "yes" s/he would like to schedule the first assessment:

Yes: May I get your telephone numbers (home and cell)? How would you prefer to be contacted? Available dates for the first assessment are [Dates] at [Times], which option would be work best with your schedule?

No: When would you like me to contact you to schedule this visit? May I get your telephone numbers (home and cell)? How would you prefer to be contacted?

Thank you.